CLINICAL TRIAL: NCT01165528
Title: Adaptive Support Ventilation vs. Conventional Ventilation Strategy in the Management of Acute Respiratory Distress Syndrome:A Randomized Controlled Trial
Brief Title: Adaptive Support Ventilation in Acute Respiratory Distress Syndrome (ARDS)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Dr. Arjun Srinivasan, senior resident, Dept of Pulmonary medicine & critical care, PGIMER
Organization: PIMERIndia (Unknown)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASVtrial
Record Dates: First submitted 2010-07-16; First posted 2010-07-20 (Estimated); Last update posted 2010-07-20 (Estimated); Status verified 2009-12

CONDITIONS: Respiration, Artificial; Respiratory Distress Syndrome, Adult
MeSH Terms: conditions — Respiratory Aspiration; Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adaptive support ventilation in ARDS (Active Comparator): patients of ARDS will be randomized to this arm to receive mechanical ventilation as per ASV protocol
  Interventions: Procedure: type of mechanical ventilation
- conventional ventilation strategy in ARDS (Active Comparator)
  Interventions: Procedure: type of mechanical ventilation

INTERVENTIONS:
Procedure: type of mechanical ventilation — patients are randomized to receive one of the two types of mechanical ventilation for ARDS

SUMMARY:
Prospective randomized controlled trial to be conducted in the Respiratory Intensive Care Unit (RICU) of Post Graduate Institute of Medical Education And Research (PGIMER),Chandigarh. The study is approved by the Institute Ethics committee. In view of lack of previous outcome data in such patients, all patients requiring RICU admission for acute respiratory distress syndrome(ARDS) between January 2010 and June 2011 are being enrolled in this pilot study.

The patients meeting the aforementioned criteria will randomly assigned to ventilation with assist control mode ventilation (ACMV group) as per the ARDSnet strategy or adaptive support ventilation (ASV group). Being the first RCT of its type, patients will be first stabilized on ACMV for 1 hour to determine the adequate minute ventilation. The randomization sequence will be computer generated. The assignments will placed in sealed opaque envelopes and each patient's assignment was made on admission to the RICU by the attending physician. Blinding of treatment is not possible.

All patients will be ventilated only by Galileo Gold ventilators (Hamilton medical systems, Bonaduz, Switzerland). Patients randomized to the ACMV group will be ventilated according to low tidal volume strategy of 6ml/kg with Fio2/PEEP as per ARDSnet table to achieve a saturation between 88-95% with the lowest possible Fio2 to maintain plateau pressures < 30 cms H2o and PH > 7.3 with option to reduce tidal volume to 4 ml/kg and increase respiratory rate to 35/ min to achieve the above said goals11.These patients will be weaned as per standard protocol of spontaneous breathing trial of 30 minutes once they are recognized eligible as per statement of the sixth International consensus conference on weaning.

DETAILED DESCRIPTION:
Inclusion criteria:

Study to include at least 40 patients admitted to RICU with diagnosis of ARDS as defined by American European consensus committee in 1994.

1. Acute onset shortness of breath(<7 days)
2. PaO2/FiO2 < 200 mm Hg (regardless of PEEP)
3. Bilateral infiltrates on frontal chest radiograph
4. <18 mm Hg when measured or no clinical evidence of left atrial hypertension

Exclusion criteria:

1. Age less than 12 years
2. Patients having underlying chronic lung disease (COPD, interstitial lung disease, pulmonary hypertension)
3. Contraindication to permissive hypercapnea (raised intracranial pressure, acute cerebrovascular disorders, acute or chronic myocardial ischemia, right ventricular failure, uncorrected severe metabolic acidosis, sickle cell anemia, tricyclic antidepressant overdose, pregnancy)

ELIGIBILITY:
Inclusion Criteria:

* Acute onset shortness of breath(<7 days)
* PaO2/FiO2 < 200 mm Hg (regardless of PEEP)
* Bilateral infiltrates on frontal chest radiograph
* <18 mm Hg when measured or no clinical evidence of left atrial hypertension

Exclusion Criteria:

* Age less than 12 years
* Patients having underlying chronic lung disease
* Contraindication to permissive hypercapnia (raised intracranial pressure, acute cerebrovascular disorders, acute or chronic myocardial ischemia, right ventricular failure, uncorrected severe metabolic acidosis, sickle cell anemia, tricyclic antidepressant overdose, pregnancy)

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-01; Primary Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Duration of mechanical ventilation | up to 4 weeks
duration of ICU stay | up to 4 weeks
duration of hospital stay | up to 8 weeks

SECONDARY OUTCOMES:
Mortality | up to 8 weeks
ease of use of ventilator mode | up to 4 weeks
frequency of blood gas analysis | up to 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Arjun srinivasan, M.D., Principal Investigator — dept of pulmonary medicine & critical care, PGIMER
Locations (1):
- Respiratory intensive care unit, PGIMER, Chandigarh, Chandigarh, India

REFERENCES:
- [Derived] Agarwal R, Srinivasan A, Aggarwal AN, Gupta D. Adaptive support ventilation for complete ventilatory support in acute respiratory distress syndrome: a pilot, randomized controlled trial. Respirology. 2013 Oct;18(7):1108-15. doi: 10.1111/resp.12126. PMID 23711230